CLINICAL TRIAL: NCT07053462
Title: Phase 1/2, Single-Arm, Open-Label Trial to Evaluate the Safety, Feasibility, and Immunogenicity of Ex Vivo CRISPR-Cas9 Gene-Edited Donor Kidneys (Knockout of HLA-A, HLA-B, and CIITA) in Human Renal Transplant Recipients
Brief Title: CRISPR-Edited HLA Donor Kidney Transplant to Reduce Rejection Risk
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AMERICAN ORGAN TRANSPLANT AND CANCER RESEARCH INSTITUTE LLC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOTCRI-101
Record Dates: First submitted 2025-06-08; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: End-Stage Renal Disease; End Stage Renal Disease on Dialysis; End Stage Renal Disease With Renal Transplant; Kidney Transplant Rejection; Kidney Tumor; Kidney Failure; Kidney Ischemia
Keywords: HLA Mismatch Immunogenicity; Transplant Rejection (Immunologic); Kidney Transplantation (Allograft); Kidney Failure; CRISPR-Cas9; Kidney Transplant; Human Leukocyte Antigen (HLA); Immunogenicity Reduction; Graft Rejection Prevention
MeSH Terms: conditions — Kidney Failure, Chronic; Carcinoma, Renal Cell; Renal Insufficiency | interventions — Kidney Transplantation; Standard of Care

STUDY DESIGN:
Intervention Model Description: Single Group Assignment (Open-Label, Non-Randomized) - All participants receive the experimental CRISPR-edited kidney transplant; there is no control arm. This is a single-arm feasibility and safety study in an early phase setting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CRISPR-Edited Donor Kidney Transplant (Experimental): All enrolled participants will receive a kidney allograft that has undergone ex vivo CRISPR-Cas9 gene editing to disrupt HLA-A and HLA-B (class I) and the CIITA gene (to broadly suppress HLA class II expression). The edited kidney is then transplanted into the patient using standard surgical techniques. Participants are maintained on a conventional post-transplant immunosuppressive regimen (with possible adjustments as appropriate for reduced graft immunogenicity). Arm description: Single-arm trial, wherein each patient is in the experimental group receiving the gene-edited kidney graft.
  Interventions: Biological: Ex Vivo CRISPR-Cas9 Gene Editing of Donor Kidney; Procedure: Kidney Transplantation with Standard Care

INTERVENTIONS:
Biological: Ex Vivo CRISPR-Cas9 Gene Editing of Donor Kidney — The donor kidney is treated outside the body with CRISPR-Cas9 ribonucleoprotein complexes targeting the genes HLA-A, HLA-B, and CIITA. This genetic intervention knocks out HLA-A/B on donor cells and disables expression of HLA-DR, -DQ, -DP by disrupting CIITA (essential for class II antigen presentation). The goal is to create a transplanted organ with greatly reduced immunogenic surface proteins. (This is a one-time genetic manipulation applied to the donor organ prior to transplantation; no direct gene therapy is given to the patient's own cells.)
Procedure: Kidney Transplantation with Standard Care — After gene editing, the donor kidney is implanted into the recipient in a surgical transplant procedure. Standard peri-operative care is provided. All patients will receive standard immunosuppressive therapy post-transplant (such as tacrolimus, mycophenolate, and prednisone, per center protocol) to prevent rejection, though the regimen may be tailored based on the edited graft's expected lower immunogenicity. Patients will be hospitalized for transplant and monitored closely during the immediate post-op period, then followed in clinic frequently for transplant aftercare.

SUMMARY:
This clinical trial investigates the transplantation of donor kidneys that have been genetically modified ex vivo using CRISPR-Cas9 genome editing to reduce immunogenicity and transplant rejection. Donor kidney grafts will have key human leukocyte antigen (HLA) genes disrupted - specifically, knockout of HLA class I heavy chains HLA-A and HLA-B, along with disabling HLA class II expression by targeting the CIITA gene (a master regulator of HLA-DR/DQ/DP). Approximately 90 adult end-stage renal disease patients will receive a CRISPR-edited donor kidney transplant. The primary objectives are to assess the safety and feasibility of this novel intervention, while secondary objectives evaluate the reduction in immune responses (immunogenicity), graft function, and the practicality of implementing ex vivo gene-edited organ transplantation in humans. By knocking out major donor HLA molecules, the trial aims to reduce T-cell and antibody-mediated recognition of the graft, potentially lowering rejection rates and reliance on high-dose immunosuppressants. Safety, including any off-target effects or unanticipated immune reactions, will be closely monitored, and transplant outcomes will be tracked for one year post-transplant.

DETAILED DESCRIPTION:
In organ transplantation, differences in HLA genes between donor and recipient are a primary driver of allorecognition and graft rejection. Mismatched donor HLA antigens are identified as "non-self" by the recipient's immune system, provoking CD8<sup>+</sup> cytotoxic T lymphocyte responses, CD4<sup>+</sup> T-helper responses, and natural killer (NK) cell activation that can damage the graft. While immunosuppressive drugs can mitigate rejection, patients remain at risk for rejection if donor HLAs are unfamiliar, and life-long immunosuppression carries significant morbidities (infection, malignancy, etc.).

Complete HLA matching is rarely achievable for all patients, especially for highly sensitized individuals with pre-formed anti-HLA antibodies. To address this, researchers have proposed rendering donor tissues "hypoimmunogenic" by removing or reducing expression of the most immunogenic HLA molecules. Preclinical studies show that eliminating key HLA class I and II antigens can prevent immune recognition and rejection of allogeneic cells. For example, genome editing of induced pluripotent stem cells to knock out HLA-A, HLA-B, and HLA-DR (via the DRA gene) successfully created universal cell grafts that evade T cell responses. Similarly, in animal models, silencing of major histocompatibility complex (MHC) genes in donor organs dramatically prolonged transplant survival. In a recent porcine study, donor lungs with reduced MHC (SLA gene) expression had markedly improved outcomes: ~71% of treated pigs survived long-term (2 years) with little to no rejection,

whereas all control pigs receiving unmodified organs rejected within 3 months. Treated animals showed reduced donor-specific antibody production and T-cell reactivity, demonstrating that lowering graft antigenicity can ameliorate rejection. These findings provide a strong rationale that knocking out donor HLA genes can reduce human allograft immunogenicity and potentially allow better graft survival with less immunosuppression.

This trial is a applying ex vivo CRISPR-Cas9 gene editing to donor organs to reduce HLA expression prior to transplantation. The editing strategy targets the donor kidney's HLA class I and II pathways: both HLA-A and HLA-B genes will be knocked out (biallelic disruption), while HLA class II expression is ablated by knocking out CIITA, a transcriptional activator required for HLA-DR, -DQ, and -DP expression. The intended result is a kidney graft largely devoid of classical HLA class I and II molecules.

Notably, HLA-C (a class I gene) may be partially retained (e.g. only one allele knocked out) to maintain a low level of class I expression - this strategy can help avoid NK cell-mediated "missing-self" responses that occur when all class I is absent. By preserving minimal HLA-C or non-polymorphic HLA-E/G expression, the graft may evade NK cell attack while still lacking the highly polymorphic HLA-A/B and class II antigens that elicit T-cell and antibody responses. The overall hypothesis is that such CRISPR-edited "stealth" kidneys will be significantly less immunogenic, leading to fewer acute rejection episodes and reduced anti-graft antibody formation, thereby improving transplant success.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age 16 to 85 years, with end-stage renal disease (ESRD) who are candidates for kidney transplantation. This includes patients on dialysis or approaching dialysis who have been evaluated and listed for transplant.
* Eligible for transplant surgery based on medical assessment (i.e., no contraindications to major surgery and transplantation). The patient's overall health status must be sufficient to undergo the transplant procedure and the required immunosuppression.
* Suitable donor organ available: A deceased-donor kidney that meets standard acceptable criteria for transplant (e.g., adequate organ function and anatomy) and is ABO blood type compatible with the recipient. The donor kidney must be allocated to the trial and available for ex vivo gene editing prior to transplantation.
* Informed consent: The patient (or legally authorized representative) is able to understand the experimental nature of the study and has voluntarily signed the informed consent form. The patient must be willing to comply with all study procedures, follow-up visits, and laboratory tests.
* Negative crossmatch (if applicable): No pre-existing anti-donor reactivity that would cause immediate graft failure. (All recipients should have a negative T and B cell crossmatch with the donor organ prior to transplant, as per standard practice, to ensure no strong baseline donor-specific antibodies, especially against any remaining donor HLA such as HLA-C.)
* Women of childbearing potential must have a negative pregnancy test and must agree to use effective contraception during the study and for a period after (to be specified, e.g., 1 year post-transplant), given the use of immunosuppressants and the unknown effects of gene-edited organ transplantation on pregnancy. Men with partners of childbearing potential should also agree to use contraception.
* High immunologic risk patients are eligible: Patients with high panel reactive antibody (PRA) levels or a history of sensitization (from prior transplants, blood transfusions, or pregnancies) are allowed and even anticipated in this trial, as the intervention is designed to benefit patients with broad HLA sensitization. For instance, patients with calculated PRA > 80% (who have difficulty finding matched donors) can be included. (Such patients must still meet the crossmatch criterion above - any existing antibodies should not target the antigens remaining on the edited graft.)
* Geographic availability: Patients must be available for long-term follow-up in the study center in China or able to travel for scheduled follow-up visits. They should be willing to remain in proximity to the transplant center for the initial post-operative period as per standard transplant care.

Exclusion Criteria:

* Active infection: Any ongoing severe infection that would contraindicate transplantation or be exacerbated by immunosuppression (e.g., active tuberculosis, untreated Hepatitis B or C, HIV with uncontrolled viremia, etc.). Patients with controlled HIV (on stable antiretroviral therapy with undetectable viral load) may be considered on a case-by-case basis, but active uncontrolled infection is excluded.
* Pregnancy or breastfeeding: Pregnant women are excluded due to the need for immunosuppressive drugs and the unknown risks of the investigational intervention on a fetus. Women who are breastfeeding are also excluded due to potential drug excretion in milk and unknown risks to the infant.
* Multi-organ transplant need: Patients requiring more than one organ transplant simultaneously (e.g., kidney + liver, or kidney + heart) are excluded, as this trial focuses on isolated kidney transplant outcomes. (A history of a prior transplant is not an automatic exclusion if the patient now only needs a kidney, but concurrent multi-organ requirements are excluded.)
* Severe co-morbidities that would significantly increase transplant risk or confound results: for example, uncontrolled cardiovascular disease (e.g., recent myocardial infarction, severe heart failure), uncontrolled diabetes with end-organ damage beyond ESRD, severe liver dysfunction, or other life-threatening illnesses unrelated to kidney failure. Such conditions could make the surgery unsafe or the outcome hard to interpret.
* Contraindications to immunosuppression: Patients with conditions that preclude standard immunosuppressive therapy (for instance, a history of anaphylaxis to tacrolimus or mycophenolate that cannot be managed, or chronic infection that would be fatally worsened by immunosuppression) are excluded. The trial still relies on baseline immunosuppressants, so patients must be able to tolerate them.
* Inability to follow the protocol: Patients with significant psychiatric disorders, cognitive impairment, or social situations that would make adherence to the study protocol and follow-up unlikely. This includes inability to give informed consent or lack of support for the intensive follow-up (for example, if the patient is incarcerated or has no fixed address, etc.).
* Prior gene therapy or organ experiment participation: Patients who have previously received any investigational gene therapy, or who have a donor-specific tolerance induction or other experimental transplant treatments ongoing, may be excluded to avoid confounding effects. (This is a precaution to attribute outcomes specifically to the CRISPR-edited organ intervention.)
* Laboratory abnormalities: Any clinically significant abnormalities in baseline labs that would pose added risk - for instance, severe leukopenia or thrombocytopenia that could worsen with immunosuppression, or uncontrolled coagulopathy that raises surgical risk.
* Donor-related exclusions: If the donor kidney, upon retrieval, is found unsuitable for gene editing or transplant (e.g., poor organ quality, unexpected disease in the organ, or if the CRISPR editing fails to achieve sufficient knockout of target genes), the transplant to that patient will not proceed under the study (the patient may either receive a standard transplant off-study or wait for another opportunity). In such a case, the patient might be withdrawn or deferred, but this is a procedural consideration rather than a characteristic of the patient.

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-18 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Related Serious Adverse Events | Day 0 to Day 365 post-transplant
  Number of participants who experience any serious adverse event (SAE) that is possibly related to the gene-edited transplant procedure within the first 12 months post-transplant.
Graft Survival at 6 Months | 6 months
  Proportion of transplanted gene-edited kidneys that remain viable and functional at 6 months post-transplant. Graft survival is defined as the kidney graft not being lost to rejection or other causes (i.e., the recipient is alive with a functioning transplant, not returning to chronic dialysis) Unit of Measure: Participants with functioning graft (n, %)

SECONDARY OUTCOMES:
Acute Rejection Episodes | 12 months
  Incidence of acute rejection events within the first 12 months post-transplant. This will be measured as the number of episodes of biopsy-confirmed acute allograft rejection (acute T-cell mediated rejection or antibody-mediated rejection) per patient, and the proportion of patients who experience at least one rejection. Unit of Measure: Episodes per participant
Donor-Specific Antibody (DSA) Development | 12 months
  Number of participants who develop de-novo anti-donor HLA antibodies (MFI ≥1000). Time Frame: Baseline to Month 12 Unit of Measure: Participants with de-novo DSA (n, %)
Mean eGFR at Month 12 | 12 months
  Average eGFR calculated by CKD-EPI at Month 12 ±7 days. Unit: mL/min/1.73 m² (mean ± SD)
Frequency of Donor-Reactive IFN-γ Producing T Cells (ELISPOT) | 12 months
  Spot-forming cells per 10⁶ PBMC in ELISPOT assay at Month 6 compared with baseline. Unit: Spot-forming cells/10⁶ PBMC (mean ± SD)
Percentage of HLA-A Alleles with Indel Mutation (NGS) | 30 days
  Indel frequency at HLA-A locus in pre-implant biopsy determined by next-gen sequencing.Unit: Percent alleles edited (%)
Overall Patient Survival at 12 Months | 12 months
  Participants alive at 12 months post-transplant.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Health Science Center (PKUHSC), Beijing, Changping, China

IPD SHARING:
Plan to Share IPD: No